CLINICAL TRIAL: NCT06899698
Title: EFFECT OF INSPIRATORY MUSCLE TRAINER ON AUTONOMIC MODULATION AND PULMONARY FUNCTION IN PATIENTS WITH STROKE
Brief Title: INSPIRATORY MUSCLE TRAINER ON AUTONOMIC MODULATION AND PULMONARY FUNCTION
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Adly A Adam (Other)
Responsible Party: Sponsor-Investigator, Adly A Adam, Lecturer of Physical Therapy, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/005300
Record Dates: First submitted 2025-03-20; First posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Hemiplegic Stroke

STUDY DESIGN:
Intervention Model Description: Brief summary; the purpose of the study is to evaluate the effect of inspiratory muscle trainer on autonomic modulation and pulmonary function in patients with stroke.
  Good evidence exists that respiratory muscle strength is significantly impaired after stroke because of decreased cortico-respiratory outflow from the damaged cortex.
  Inspiratory muscle training (IMT) improves the interplay of the respiratory pump, hemodynamic, cerebrovascular and postural balance responses.
  Sixty chronic hemiplegic patients will be randomly allocated into; Study group will receive IMT, their medications in addition to the traditional training for eight weeks; Control group will receive their medications in addition to the traditional training for eight weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Study Group (Experimental): Thirty chronic hemiplegic patients with mild cognitive impairment, and suffering from orthostatic hypotension will receive inspiratory muscle training for 30 minutes per day for at least 3 days a week for 8 weeks, medications, and traditional training along 8 weeks.
  Interventions: Other: Inspiratory muscle training; Other: Traditional Training
- Control Group (Other): Thirty chronic hemiplegic patients with mild cognitive impairment, and suffering from orthostatic hypotension will receive their medications, and traditional training along 8 weeks.
  Interventions: Other: Traditional Training

INTERVENTIONS:
Other: Inspiratory muscle training — Only participants in the Study group 'Thirty chronic hemiplegic patients with mild cognitive impairment, and suffering from orthostatic hypotension' will receive inspiratory muscle training using Respiratory muscle strength: Threshold Inspiratory muscle trainer (TIMT): Philips Respironics model (Tayland- B00J417PHM), for 30 minutes per day for at least 3 days a week for 8 weeks.
  Arms: Study Group
Other: Traditional Training — Both the study and control group 'Sixty chronic hemiplegic patients with mild cognitive impairment, and suffering from orthostatic hypotension' will receive a. bobath technique 'passive mobilization associated with tactile and proprioceptive stimuli aims to inhibits spasticity'; b. Proprioceptive neuromuscular facilitation 'based on spiral and diagonal patterns of movements in line to achieve normal movements' c. Rood technique 'focuses on the developmental sequence of recovery (from basic to complex) and the use of sensory stimulation to facilitate movement and postural responses' d. Johnstone method 'includes positioning and splinting to inhibit abnormal patterns and controlling tone to restore central control' e. Functional electrical stimulation; f. Balance training, j. Pelvic, and gait training, h. Activities of daily living, and finally, g. Sensrimotor training 'Active and active-assistive range-of motion exercises, Graded activities Start with easy activities'.

SUMMARY:
Stroke individuals with hemiplegia often display difficulties in mobility, cardiopulmonary function...etc. All stroke patients had restrictive pulmonary dysfunction. Therefore, respiratory training improves their respiratory capacity, and orthostatic stress mediated respiratory, cardiovascular and autonomic response. Respiratory muscle training interventions are efficient in terms of pulmonary functional parameters. In advanced line, this study will be conducted to evaluate inspiratory muscle trainer effect on autonomic modulation and pulmonary function in stroke patients.

DETAILED DESCRIPTION:
The second trigger of death and the most frequent life-threatening neurological disease are now strokes. Stroke is the third main cause of the death & disability in Egypt. According to world health organization; from the total world's population, nearly 18.6 had severe disability and 79.7 million had moderate long-term disability. Respiratory dysfunction is a common complication of stroke, with an incidence of over 60%. Despite the high prevalence of stroke-induced respiratory dysfunction, how disordered breathing influences recovery and cognitive outcomes after ischemic stroke is unknown.

Patients with hemiplegia exhibited diminished respiratory muscle strength and pulmonary function at a more severe motor dysfunction level. Impaired inspiratory muscle strength was associated with reduced balance ability and limitations in activities required for daily living.

in the same line this study will be conducted to find out the effect of inspiratory muscle trainer on autonomic modulation and pulmonary function in patients with stroke.

Sixty chronic hemiplegic patients who aged from 55:65 years old will be recruited, and randomly divided into 2 equal groups; study group will receive threshold inspiratory muscle trainer for 8 weeks (24 sessions) and their medications, and traditional training, where control group will receive their prescribed medications in addition to the same traditional training.

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemiplegic post stroke patients 'at least 6months'
* Men.
* Age ranged 55-65years old.
* Body mass index ranged from 29.9- 34.9 kg/m2
* Mini-Mental State Examination (MMSE) scores of 23-27 indicate mild cognitive impairment
* Did not participate in any selective exercise program for the respiratory muscles before.
* Participants suffering from orthostatic hypotension a systolic BP decline ≥20 mm Hg or a diastolic BP decline ≥10 mm Hg on position change from sitting to standing.

  * Smokers will be defined as those (who had smoked >400 cigarettes in their lifetime)

Exclusion Criteria:

* Unstable cardiovascular problems.
* Asthmatic patient.
* Implanted pacemaker
* Patients with chest infection.
* Patients with pleural diseases.
* Primary valvular disease.
* History of spontaneous pneumothorax.
* Clinically significant peripheral vascular disease.
* Severe anemia being unable to follow RMT instructions or complete the questionnaires of the study due to cognitive impairment .
* Previous lung surgery.
* Long-term oxygen treatment.
* Patients with chronic renal failure.
* Any patient enrolled in an anther research study for at least 30 days.
* Facial affection

Ages: 55 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men; their age range 55-65 years old suffering from chronic hemiplegic patients, their BMI ranged from 29.9- 34.9 kg/m2 , also with mild cognitive impairment
Enrollment: 60 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure | Pre-treatment, and Post-treatment of the 8-weeks of the study protocol (24 Sessions).
  systolic, diastolic blood pressure and mean arterial blood pressure those will be measure using Mercury sphygmomanometer and stethoscope (China ,1600G004).
Pulmonary Function test | Pre-treatment, and Post-treatment of the 8-weeks of the study protocol (24 Sessions).
  Pulmonary function test using Spirometry will be used to evaluate (Compact; Vitalograph; Buckingham, England) FVC, FEV1, FEV1 / FVC will be measured three times per each time of evaluation on a computerized spirometer

SECONDARY OUTCOMES:
Functional capacity and orthostatic hypotension assessment | Pre-treatment, and Post-treatment of the 8-weeks of the study protocol (24 Sessions).
  Sit to stand test will be used for functional capacity assessment in addition to assessing the blood pressure from sitting to standing positions before and after treatment
Cognitive function | Pre-treatment, and Post-treatment of the 8-weeks of the study protocol (24 Sessions).
  Cognitive function will be assessed using the Mini-Mental State Examination (MMSE) scores that is a tool that can be used to systematically and thoroughly assess mental status. It is an 11-question measure that tests five areas of cognitive function: orientation, registration, attention and calculation, recall, and language. The maximum score is 30. A score of 23 or lower is indicative of cognitive impairment. The MMSE takes only 5-10 minutes to administer and is therefore practical to use repeatedly and routinely.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Mohamed Ahmed, Bachelor of Physical Therapy, Principal Investigator — Physical Therapy Faculty; Ebtesam Nabil Abdel Mohsen, Lecturer of Physical Therapy, Study Director — Physical Therapy Faculty; Ebtesam Mohamed Fahmy, Professor of Neurology, Study Director — faculty of medicine; Zeinab Mohamed Helmy, Professor of Physical Therapy, Study Chair — faculty of physical therapy
Locations (1):
- Physical Therapy Faculty, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No